CLINICAL TRIAL: NCT03094494
Title: Double Carbapenem as Rescue Strategy for the Treatment of Severe Carbapenemase-Producing Klebsiella Pneumoniae Infections: A Two-Center Matched Case-Control Study
Brief Title: Double Carbapenem as Rescue Strategy for the Treatment of Carbapenemase-Producing Klebsiella Pneumoniae Infections
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Gennaro De Pascale, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: UCSC14669/15 359/2015
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Carbapenem; Klebsiella Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Double Carbapenem Group: Patients underwent Double carbapenem treatment
  Interventions: Other: none intervention
- Standard Treatment Group: Patients who were not treated with the double carbapenem
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — none intervention

SUMMARY:
An observational two-center case-control study exploring the clinical impact of double-carbapenem use in a population of critically il patients with severe carbapenem-resistant Klebsiella pneumoniae infection

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. ICU admission between November 2012 and December 2015;
3. documented CR-Kp invasive infection;
4. targeted antibiotic therapy lasting ≥ 72 hours

Exclusion Criteria

1. Klebsiella infection, susceptible to carbapenems
2. Duration of antimicrobial therapy less than 72 hours
3. Data not completely available from the electronically medical chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with severe CR-Kp infection
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 day
  mortality after 28 day from infection

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] De Pascale G, Martucci G, Montini L, Panarello G, Cutuli SL, Di Carlo D, Di Gravio V, Di Stefano R, Capitanio G, Vallecoccia MS, Polidori P, Spanu T, Arcadipane A, Antonelli M. Double carbapenem as a rescue strategy for the treatment of severe carbapenemase-producing Klebsiella pneumoniae infections: a two-center, matched case-control study. Crit Care. 2017 Jul 5;21(1):173. doi: 10.1186/s13054-017-1769-z. PMID 28679413